CLINICAL TRIAL: NCT04546802
Title: Open Label Trial to Study the Efficacy and Safety of MK-5172 and MK-8742 +/- Ribavirin (RBV) in the Treatment of Hepatitis C G1 and 4, in Patients Eligible for Liver Transplant (HCC) or Curative Therapy or Clinically Stable Disease Post Local Resection, Embolization or Ablative Therapy
Brief Title: HepATocellular Cancer Hcv Therapy Study
Acronym: HATCHeT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment will be too difficult due to available PBS funded treatment and recent Australian clinical guidelines will conflict with the premise of the study.
Sponsor: Bayside Health (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Austin Hospital, Melbourne Australia (Other)
Responsible Party: Principal Investigator, Ms. Rowan Frew, Manager Research and Ethics Department, Bayside Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 288/18
Record Dates: First submitted 2018-10-14; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Liver Cell Carcinoma; Hepatitis C
Keywords: hepatitis C; Elbasvir/grazoprevir; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Active Comparator): This group will undergo immediate treatment of the HCV once HCC complete response (CR) has been confirmed
  Interventions: Drug: Elbasvir / Grazoprevir Oral Tablet
- Delayed treatment (Active Comparator): This group will delay commencement of the HCV treatment until 6 months after HCC complete response (CR) has been confirmed
  Interventions: Drug: Elbasvir / Grazoprevir Oral Tablet

INTERVENTIONS:
Drug: Elbasvir / Grazoprevir Oral Tablet — Elbasvir / Grazoprevir

SUMMARY:
Subjects with Hepatitis C Virus (HCV) infection, genotype 1 or 4 and with hepatocellular carcinoma (HCC) and a complete response to HCC therapy will be randomised to immediate or delayed (6 months) HCV therapy with Elbasvir (MK-8742) and Grazoprevir (MK-5172) [EBR/GZR].

DETAILED DESCRIPTION:
Two cohorts (A and B) of patients with chronic HCV infection will be enrolled. Patients will be eligible for enrollment if they fulfill the study inclusion and exclusion criteria and have achieved a complete tumour response (CR) 3 months (+/- 14 days) following HCC treatment

* Cohort A: Patients with Barcelona Clinic Liver Cancer (BCLC) stage 0 or A HCC who have received curative therapy defined as either; liver transplantation, surgical resection or local ablation with curative intent and attained a radiologically confirmed CR. (N=50)
* Cohort B: Patients who are non-eligible for curative therapy but have attained a radiologically confirmed CR. post embolization or ablative therapy and have chronic HCV infection. (N=50) Given the existing uncertainty regarding the impact of direct acting antiviral (DAA) therapy on HCC recurrence, study participants will be randomized to receive DAA treatment as "immediate" ie upon study enrollment or "delayed" ie treatment commenced ≥ 6months following documentation of complete response based on radiological assessment indicating no residual arterial enhancing disease..

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C diagnosed as the HCV RNA (≥ 10,000 IU/mL in peripheral blood) at the time of screening
* Genotype inclusions
* Have documented chronic HCV GT1 or GT4, (with no evidence of nontypeable or mixed genotype) infection
* HCC diagnosed on the basis of histology or according to AASLD radiological criteria,
* Written informed consent granted prior to initiation of any study-specific screening procedures
* Patients aged 18 to 70 years-old;
* Child-Pugh ≤≤ A6
* BCLC stage 0, A HCC or no detectable HCC in a patient who has undergone a curative form of treatment (liver transplantation, surgical resection of local ablative therapy with curative intent) OR BCLC-B disease but clinically stable with non-evidence of disease progression as demonstrated by either Triphasic CT or contrast MRI at least 3 months after the last HCC treatment.

Exclusion Criteria:

* Enrolment in other investigation / experimental therapies

  * Prior or current use of Sorafenib or other systemic chemotherapy
  * Life expectancy < 12 months (unless transplantation eligible)
  * Unable to provide informed consent
  * Previous or concurrent cancer that is distinct from HCC in primary site or histology, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, and superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to enrollment is permitted.
* Any condition that in the opinion of the investigator would impair participation in the trial.
* Coinfected with human immunodeficiency virus (HIV) infection or Hepatitis B virus (e.g. HBsAg positive).
* History of congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification within 6 months prior to study entry; active coronary artery disease (CAD); clinically significant bradycardia or other uncontrolled, cardiac arrhythmia defined as ≥ Grade 3 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, or uncontrolled hypertension; myocardial infarction occurring within 6 months prior to study entry (myocardial infarction occurring > 6 months prior to study entry is permitted)
* Active clinically serious infections defined as ≥ Grade 3 according to NCI CTCAE, version 4.03 6. Any medical, psychological, or social conditions, particularly if unstable, including substance abuse, that may, in the opinion of the Investigator, interfere with the subject's safety or participation in the study, protocol compliance, or evaluation of the study results
* Concomitant interferon therapy or therapies for active Hepatitis C Virus (HCV) infection. Prior interferon and/or ribavirin therapy is not a contraindication to enrolment however previous treatment with direct acting antiviral treatment is an exclusion
* Pregnancy or breast-feeding
* Inability to swallow oral medications
* Clinically significant gastrointestinal bleeding occurring ≤ 3 months prior to study entry or Large gastric-esophageal varices (larger than 5 cm) or previous history of gastric-esophageal bleeding due to varices.
* Fulfills exclusion criteria on biochemistry results:

  * Creatinine Clearance <50 mL/min
  * Hemoglobin <11 g/dL for females and <12 g/dL for males
  * Platelets <75 x 103/μL
  * Serum Albumin < 3.0 g/dL
  * INR >1.7
  * HbA1c >10%
  * ALT >10XULN, AST >10XULNtherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Viral eradication | 12 weeks
  Eradication of Hepatitis C virus determined by undetectable viral load

SECONDARY OUTCOMES:
HCC recurrence rate following HCC treatment | 6 and 12 month
  impact of DAA therapy on 6 and 12 month HCC recurrence rate following HCC treatment
Recurrence free survival | 5 years
  Recurrence free survival
Disease free survival | 5 years
  Disease free survival
Time to HCC recurrence / progression | 5 years
  Time to HCC recurrence / progression
Adverse events | Up to 5 years
  Safety and tolerability of Elbasvir/grazoprevir determined by adverse events

OTHER OUTCOMES:
Overall survival | Up to 5 years
  Overall survival determined by proportion surviving

CONTACTS AND LOCATIONS:
Overall Officials: William kemp, MBBSFRACPPhD, Principal Investigator — The Alfred

IPD SHARING:
Plan to Share IPD: No